CLINICAL TRIAL: NCT06935136
Title: A Single-Arm, Multicenter, Open-Label Clinical Study to Evaluate the Efficacy and Safety of Axicabtagene Ciloleucel Injection as First-Line Therapy of High-Risk Large B-Cell Lymphoma
Brief Title: Study to Evaluate the Efficacy and Safety of Axicabtagene Ciloleucel Injection as First-Line Therapy of High-Risk Large B-Cell Lymphoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Ruijin Hospital, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RJ-1L HR-01
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: CAR-T Cell Therapy; High-risk Large B-cell Lymphoma (LBCL)
Keywords: axi-cel; car-t; LBCL
MeSH Terms: interventions — axicabtagene ciloleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group (Experimental): Participants will receive cyclophosphamide 500 mg/m^2/day intravenously (IV) and fludarabine 30 mg/m^2/day IV conditioning chemotherapy for 3 days followed by axicabtagene ciloleucel（Axi-cel） administered as a single IV infusion at a target dose of 2 x 10^6 anti-cluster of differentiation (CD)19 chimeric antigen receptor (CAR) transduced autologous T cells/kg on Day 0.
  Interventions: Drug: Axicabtagene Ciloleucel

INTERVENTIONS:
Drug: Axicabtagene Ciloleucel — A single infusion of chimeric antigen receptor (CAR)-transduced autologous T cells
  Other Names: FKC-876; Axi-cel

SUMMARY:
The goal of this is Single-Arm, Multicenter, Open-Label Clinical Study is to Evaluate the Efficacy and Safety of Axicabtagene Ciloleucel Injection(Axi-cel) as First-Line Therapy of High-Risk Large B-Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed LBCL (Large B-Cell Lymphoma) according to the WHO 2016 classification, including the following subtypes:DLBCL-NOS (Diffuse Large B-Cell Lymphoma, Not Otherwise Specified),HGBL (High-Grade B-Cell Lymphoma, including HGBL with MYC, BCL-2, and/or BCL-6 rearrangements (DHL/THL), HGBL-NOS),DLBCL transformed from follicular or marginal zone lymphoma, eligible if the patient has not previously received anthracycline-containing therapy
* International Prognostic Index (IPI) score of 2-5 at initial diagnosis.
* Individuals must have a positive interim positron emission tomography (PET) (Deauville PET score of 4 or 5) after 2 cycles (PET2+) of chemoimmunotherapy or high-risk ctDNA status (ctDNA levels not reduced by at least 2-log after two cycles of R-chemotherapy)
* Age of 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Adequate renal, hepatic, pulmonary, and cardiac function, defined as:

  * Creatinine clearance (estimated by Cockcroft-Gault formula) ≥ 60 mL/min
  * Serum ALT/AST ≤ 2.5 × Upper Limit of Normal (ULN)
  * Total bilirubin ≤ 1.5 × ULN (except for patients with Gilbert's syndrome)
  * Left ventricular ejection fraction ≥ 50%, no pericardial effusion as determined by echocardiography, and no clinically significant arrhythmias No clinically significant pleural effusion
  * Baseline peripheral oxygen saturation > 92% under room air ventilation
  * At least one measurable lesion.
  * For women of childbearing potential, a negative serum pregnancy test is required (women who have undergone surgical sterilization or are postmenopausal for at least 2 years are considered not to be of childbearing potential).

Exclusion Criteria:

* According to the WHO 2016 classification, patients with the following subtypes are excluded:

  * LBCL with T-cell/histiocyte-rich background
  * Primary central nervous system DLBCL
  * PMBCL (Primary Mediastinal B-Cell Lymphoma)
  * B-cell lymphoma, unclassifiable, with features intermediate between DLBCL and classical HL (Hodgkin Lymphoma)
  * Burkitt lymphoma
  * History of Richter transformation in chronic lymphocytic leukemia
* Presence of detectable malignant cells in the CSF (cerebrospinal fluid), brain metastases, or history of central nervous system involvement by lymphoma.

Presence of cardiac involvement by lymphoma.

* Prior treatment for LBCL other than two cycles of R-chemotherapy.
* History of severe immediate hypersensitivity reaction to any of the drugs used in this study.
* Presence of central nervous system disorders: history of stroke, transient ischemic attack, or reversible posterior leukoencephalopathy syndrome (PRES) within 12 months prior to enrollment.
* History of acute or chronic active hepatitis B or C infection, unless HBV-DNA and HCV-RNA levels are below the level of detection.
* Human immunodeficiency virus (HIV) positivity, unless on appropriate antiretroviral therapy with undetectable viral load by PCR and a CD4 count > 200 cells/µL.
* Any medical condition that may interfere with the assessment of the safety or efficacy of the study treatment.
* History of clinically significant cardiac disease within 12 months prior to enrollment.
* Any other condition deemed by the investigator as unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-10-09 (Estimated); Study Completion 2028-04-09 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate Per the Lugano Classification as Determined by Study Investigators | Up to 2 years
  CR Rate is the percentage of participants with CR (complete metabolic response (CMR); complete radiological response (CRR)). CMR: positron emission tomography (PET) 5-point scale (5-PS) scores of 1 (no uptake above background), 2 (uptake ≤ mediastinum), 3 (uptake > mediastinum but ≤ liver) with/without a residual mass); no new lesions; and no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow (BM). CRR: target nodes/nodal masses regressed to ≤ 1.5 cm in longest transverse diameter of lesion (LDi); no extralymphatic sites of disease; absent non-measured lesion (NMLs); organ enlargement regress to normal; no new sites; and bone marrow normal by morphology.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per the Lugano Classification as Determined by Study Investigators | Up to 2 years
  ORR: percentage of participants with CR (CMR;CRR) or PR (partial metabolic response (PMR); partial radiologic response (PRR)). CMR: PET 5PS scores of 1 (no uptake above background, 2 (uptake ≤mediastinum), 3 (uptake >mediastinum but ≤liver) with/without a residual mass; no new lesions; no evidence of FDG-avid disease in BM. CRR: target nodes/nodal masses regressed to ≤1.5 cm in LDi; no extralymphatic sites of disease; absent NMLs; organ enlargement regress to normal; no new sites; bone marrow morphology normal. PMR: scores 4 (uptake moderately >liver),5 (uptake markedly >liver, new lesions) with reduced uptake compared with baseline and residual mass; no new lesions; responding disease at interim/residual disease at end of treatment (EOT). PRR: ≥50% decrease in sum of the product of perpendicular diameters (SPD) of up to 6 target measurable nodes and extra-nodal sites; absent/normal, regressed, but no increase of NMLs; spleen regressed by >50% in length beyond normal; no new sites.
Complete Metabolic Response (CMR) - determined by investigator | 3 months from axi-cel infusion
  CMR from axi-cel infusion (without additional anticancer therapy) based on investigator disease assessment according to PET-scan (using the Lugano Response Criteria)
Duration of Response (DOR) Per the Lugano Classification | Up to 2 years
  DOR is defined only for participants who experience an objective response after axicabtagene ciloleucel infusion and is the time from the first objective response to disease progression (PD) (Lugano classification) or death from any cause. Objective response is defined in outcome measure (OM) 2. PD is defined as a score 4 (uptake moderately > liver) or 5 (uptake markedly >liver and/or new lesions) with an increase in intensity of uptake from baseline; new FDG-avid foci consistent with lymphoma at interim or end of treatment assessment; new FDG-avid foci consistent with lymphoma rather than another etiology (eg, infection, inflammation); new or recurrent FDG-avid foci in bone marrow. Kaplan-Meier (KM) estimates were used for analysis.
Progression-Free Survival (PFS) | Up to 2 years
  PFS was defined as the time from axicabtagene ciloleucel infusion date to the date of disease progression per Lugano classification or death from any cause.
Overall Survival (OS) | Up to 2 years
  OS is defined as the time from axicabtagene ciloleucel infusion to the date of death from any cause.
Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (SAE) | Up to 2 years
  An AE was any untoward medical occurrence in a participant in a clinical trial participant, which did not necessarily have a causal relationship with the treatment. Treatment-emergent adverse events were defined as any adverse event with onset on or after the axicabtagene ciloleucel infusion. Serious adverse event was defined as an event that resulted in the following: death; life-threatening situation; in-patient hospitalization or prolongation of existing hospitalization; persistent or significant disability or incapacity; congenital anomaly or birth defect; and medically important event or reaction.

OTHER OUTCOMES:
Peak Serum Level of Granzyme B, Interferon-gamma (IFNg), Interleukin (IL)-2, IL-5, IL-6, IL-8 | Up to Week 4
  Peak is defined as the maximum post-baseline level of cytokine from baseline to Week 4.
Peak Serum Level of C-Reactive Protein (CRP) | Up to Week 4
  Peak is defined as the maximum post-baseline level of cytokine from baseline to Week 4.
Peak Serum Level of Ferritin | Up to Week 4
  Peak is defined as the maximum post-baseline level of cytokine from baseline to Week 4
Proportion of participants experiencing a clinically meaningful improvement in physical functioning and fatigue (EORTC QLQ-C30) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- China, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No